CLINICAL TRIAL: NCT06944743
Title: Predictors of Improvement Afetr Trasurtheral Resection of Prostate in Patients With Underactive Bladder and Bladder Outlet Obstruction
Brief Title: TURP Inpatient With Underactive Bladder With BOO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Emad Abdellah Ali Mostafa, Director,Head of urology,Principal investigator,clinical professor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soh-Med-25-3__IMD
Record Dates: First submitted 2025-03-23; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: TURP Syndrome; Retention, Urinary; Prostate Disease
MeSH Terms: conditions — Urinary Retention; Prostatic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transurtheral Resection of prostate in underactive bladder with bladder outlet obstruction (Other): TURP involves an endoscopic approach via the patient's urethra to surgically remove the inner portion of the prostate that encircles the urethra. A bipolar electrified wire loop is used to remove the portion of the prostate between the bladder neck and the verumontanum to a depth of the surgical capsule. Before the resection is begun, the bladder should be inspected for any bladder pathology (e.g., tumor, diverticula or stones).
  The bladder neck, trigone, and position of the ureteral orifices, verumontanum, and external sphincter should be noted. Three-way Foley catheter is usually placed to and traction for a short time, release of traction based on clearance of hematuria.
  Interventions: Procedure: Transurtheral Resection of prostate ( TURP)

INTERVENTIONS:
Procedure: Transurtheral Resection of prostate ( TURP) — TURP involves an endoscopic approach via the patient's urethra to surgically remove the inner portion of the prostate that encircles the urethra. A bipolar electrified wire loop is used to remove the portion of the prostate between the bladder neck and the verumontanum to a depth of the surgical capsule. Before the resection is begun, the bladder should be inspected for any bladder pathology (e.g., tumor, diverticula or stones).
  The bladder neck, trigone, and position of the ureteral orifices, verumontanum, and external sphincter should be noted. Three-way Foley catheter is usually placed to and traction for a short time, release of traction based on clearance of hematuria.

SUMMARY:
The study is for aproved that Transurtheral Resection of prostate is good for patient with underactive bladder or not.

DETAILED DESCRIPTION:
Introduction:

Aging men frequently develop lower urinary tract symptoms (LUTS). These symptoms are commonly attributed to bladder outlet obstruction by benign prostatic hyperplasia (BPH) and the clinical condition is termed BPH. However, recent studies have implicated many factors in the pathogenesis of LUTS in addition to BPH. These include prostate inflammation and fibrosis, increased serum estrogen/testosterone ratio, diabetes, the metabolic syndrome, sleep apnea, polyuria and changes in bladder function .

Transurethral resection of prostate (TURP) is a time-tested gold standard surgical option for dealing with LUTS in men having benign prostatic enlargement (BPE) . Persistence of LUTS is reported in 5%-35% of patients undergoing TURP .

Detrusor Under activity (DUA) is defined by the International Continence Society (ICS) as "a contraction of reduced strength and/or duration, resulting in prolonged bladder emptying and/or failure to achieve complete bladder emptying within a normal time span" . Detrusor underactivity was demonstrated in 17% men presenting with LUTS after urodynamic evaluation .

Male DUA definition remains controversial and no effective treatment is consolidated. The role of prostatic surgery in male DUA is not clear. The primary endpoint was the clinical and voiding improvement based on International Prostate Symptom Score (IPSS) and the maximum flow rate in uroflowmetry (Qmax) within 12 months.

DUA is a common association for persistence of symptoms after TURP in such patients .

Projected isovolumetric pressure (PIP) was proposed by Schäfer, who used a straight line to represent the Bladder Outlet Relation (BOR) and then "projected" back to the y-axis (pdet) from the point representing pdet@Qmax to obtain the isovolumetric pressure. This projection is calculated by the formula PIP = Pdet@Qmax + KQmax where K is a fixed constant representing the steepness of the angle of the BOR to x-a axis .

K is dependent on the specific population studied and differs between men and women .In men it is usually taken as 5. The suggested groupings for PIP are as follows:

* >150 - strong contractility
* 100 to 150 - normal contractility
* 50 to 100 - weak contractility
* <50 - very weak contractility Surgical failure is more likely to occur in patients with detrusor dysfunction and lower baseline Bladder outlet obstruction index (BOOI ). It has also been found that the degree of preoperative BOO is positively associated with improvement and QoL after TURP . Therefore, a preoperative Pressure Flow Study (PFS) is recommended for optimal selection of patients who are more suitable for surgery by measuring BOOI and assessing detrusor function. BOOI (PdetQmax-2Qmax) .

Conflicting results create dilemma about the efficacy and results of TURP in patients with BPE and bladder underactivity . In this study, Investigators evaluate the Predictors of Improvement after Transurethral Resection of Prostate in Patients with Underactive Bladder and Bladder outlet obstruction.

Aim of the work:

To pick up the predictors of improvement after Transurethral Resection of Prostate in Patients with Underactive Bladder and Bladder outlet obstruction.

Pre-Operative Predictors:

1. Age.
2. Body mass index.
3. pre-operative urinary flow rate.
4. International Prostate Symptom Score (IPSS).
5. Urodynamic parameters (BCI, BOOI, PVR and bladder capacity……...etc.).
6. Prostate size.
7. Degree of vesicoureteral reflux (if present).
8. Functional Bladder Capacity.

Intra-Operative Predictors:

1. Surgical technique.
2. Prostatic Resected weight.
3. Intra-operative complications.
4. Prostate type (Bilobular,trilobular,adenomatous or fibrous).
5. TURP syndrome.

Post-Operative Predictors:

1. Catheterization duration.
2. post-operative urinary retention.
3. Complications: (e.g., infections, stricture).
4. Early post-operative voiding trials.
5. Measure degree of vesicoureteral reflux after TURP.
6. Functional bladder Capacity after TURP.

Urodynamic Predictors:

1. Detrusor contractility.
2. Bladder outlet obstruction.
3. Functional bladder capacity.
4. UAB severity: Mild/moderate (UAB symptoms).
5. Maximum urinary flow rate.
6. Compliance of bladder.

Other Predictors:

1. Patient expectations: Realistic expectations and mental health influence.
2. Co-morbidities.
3. pre-operative physical therapy.
4. Smoking cessation.

Surgical Technique:

Perioperative antibiotic coverage for surgery should be carefully considered especially for patient who has an indwelling catheter (urethral or suprapubic).

TURP is performed using spinal anesthesia. TURP involves an endoscopic approach via the patient's urethra to surgically remove the inner portion of the prostate that encircles the urethra. A bipolar electrified wire loop is used to remove the portion of the prostate between the bladder neck and the verumontanum to a depth of the surgical capsule. Before the resection is begun, the bladder should be inspected for any bladder pathology (e.g., tumor, diverticula or stones).

The bladder neck, trigone, and position of the ureteral orifices, verumontanum, and external sphincter should be noted. Three-way Foley catheter is usually placed to and traction for a short time, release of traction based on clearance of hematuria.

In the absence of significant capsular perforation or persistent bleeding, the catheter can be removed after 24 to 48 hours.

.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with BOO and UAB
* Age ≥ 40 years.

Exclusion Criteria:

* Patient insulin dependent diabetes
* Patient with history of cerbrovascular stroke or hemarrage.
* History of prior prostate surgery.
* Urethral pathology or surgery.
* Patient with prostate or bladder cancer.
* Spinal and pelvic trauma or surgery.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in international prostate symptome score (IPSS) score. | 3 month .
  Outcome measure Detrusar pressure at maximum flow (Pdet-Qmax unit:CmH2O)

CONTACTS AND LOCATIONS:
Overall Officials: Emad Mostafa, MD, Principal Investigator — Assistant lecture
Locations (1):
- Emad Abdellah Ali Mostafa, Sohag, Egypt